CLINICAL TRIAL: NCT05201820
Title: Cryoanalgesia for Pain Management After Pectus Excavatum Repair. COPPER Study (CryoanalgesiafOr Pain Management After Pectus Excavatum Repair): a Randomized Controlled Trial
Brief Title: Cryoanalgesia for Pain Management After Pectus Excavatum Repair
Acronym: COPPER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Giannina Gaslini (Other)
Responsible Party: Principal Investigator, Nicola Disma, MD, Head of Research and Innovation Unit, Istituto Giannina Gaslini
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COPPER
Record Dates: First submitted 2021-09-20; First posted 2022-01-21 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Pectus Excavatum
MeSH Terms: conditions — Funnel Chest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care (No Intervention): Epidural analgesia
- Cryoanalgesia (Experimental): Cryoanalgesia
  Interventions: Device: Cryoanalgesia

INTERVENTIONS:
Device: Cryoanalgesia — Cryoanalgesia will be applied during surgery on 6 intercostal nerves each side
  Arms: Cryoanalgesia

SUMMARY:
Cryoanalgesia for pain management after pectus excavatum repair. COPPER study (CryoanalgesiafOr Pain management after Pectus Excavatum Repair): a randomized controlled trial.

Determine if, in patients more than 12 years of age having cryoanalgesia for pectus excavatum repair analgesia improves the standard of care (epidural analgesia) in term of pain relief and return to normal life 2 weeks after surgery.

Randomized active controlled, parallel group, single-centre, trial (category IIb medical device).

88 patients aged more than 12 years of age scheduled for pectus excavatum repair. After randomization, patients will receive intraoperative cryo-analgesia or standard of care (epidural-analgesia).

PedsQLscale (23 items) two weeks after surgery.

Patients will be followed for 6 months after surgery to determine time until return to normal life and occurrence of any complication related to the use of cryo-analgesia. Numeric Rating Scale (NRS), CALI9, YAPFAQ will be measured at fixed times to determine pain intensity and limitations due to pain. Risk factors for prolonged pain and time needed until achieving discharge criteria from hospital will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing pectus excavatum repair with NUSS technique
* aged 12 years or above12
* informed consent signed for cryoanalgesia

Exclusion Criteria:

- Age of 11 years or below

* Refuse to receive cryoanalgesia or epidural catheter as primary pain relief
* Any contraindication to cryoanalgesia
* Difficult follow-up for geographical reasons and/or impossibility by the patient to understand how to perform self-measurements

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-03-19 (Actual); Study Completion 2024-03-19 (Actual)

PRIMARY OUTCOMES:
Quality of Life by PedsQL 23 items | Two weeks after surgery
  Quality of life after surgery

SECONDARY OUTCOMES:
YAPFAQ (Youth Acute Pain Functional Ability Questionnaire) | One week after surgery
  A scale for assessment of activity limitations in children and adolescents. Range fro 0 to 100
Pain by VAS | 1-14 days after surgery
  Numeric pain score 0-10
Thoracic hypo-aesthesia | Six months after surgery
  Cold test assessment (Yes/No)

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Giannina Gaslini, Genova, Italy

IPD SHARING:
Plan to Share IPD: Yes
Once final publication is accepted, other researchers can request IPD
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: At the time of submission for publication
Access Criteria: By request

REFERENCES:
- [Background] Arshad SA, Hatton GE, Ferguson DM, Li LT, Austin MT, Tsao K; PAPS SPONSOR. Cryoanalgesia enhances recovery from minimally invasive repair of pectus excavatum resulting in reduced length of stay: A case-matched analysis of NSQIP-Pediatric patients. J Pediatr Surg. 2021 Jul;56(7):1099-1102. doi: 10.1016/j.jpedsurg.2021.03.017. Epub 2021 Mar 24. PMID 33853733
- [Derived] Bastianello M, Torre M, Bonfiglio R, Calevo MG, Palomba L, Uva P, Kanapari A, Lorenzoni G, Disma N; COPPER consortium. Cryoanalgesia for Pain Management After Pectus Excavatum Repair (COPPER) in Adolescents: A Randomized Controlled Trial. Paediatr Anaesth. 2025 May;35(5):347-358. doi: 10.1111/pan.15090. Epub 2025 Mar 4. PMID 40035332